CLINICAL TRIAL: NCT04930991
Title: A Phase 0 Study of High Dose Omeprazole in Patients With Pancreatic Cancer Planning to Undergo Surgical Therapy for Evaluating Changes of Biomarkers
Brief Title: High Dose Omeprazole in Patients With Pancreatic Cancer
Acronym: OU202005AJ
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OU-SCC-Omeprazole
Record Dates: First submitted 2021-03-29; First posted 2021-06-18 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Exocrine Pancreatic Cancer
Keywords: pancreatic cancer; omeprazole
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A (High Dose) (Experimental): Omeprazole, 80 mg, PO, BID for 12-14 days prior to surgical therapy of pancreatectomy. All 30 subjects in Arm A to be enrolled prior to Arm B cohort enrollment.
  Interventions: Drug: Omeprazole
- Arm B (Normal Dose) (Placebo Comparator): Omeprazole, 20 mg, PO, QD for 12-14 days prior to surgical therapy of pancreatectomy.
  Interventions: Drug: Omeprazole

INTERVENTIONS:
Drug: Omeprazole — Treatment will consist of Omeprazole 12-14 days prior to surgical therapy of pancreatectomy.

SUMMARY:
The purpose of this study is to test the safety of high dose omeprazole and see what effects that it has on patients with exocrine pancreatic cancer.

DETAILED DESCRIPTION:
During this study patients will receive treatment of omeprazole at the dose depending on group enrollment

* Group A will receive omeprazole 80 mg, twice a day for 12-14 days unless unacceptable toxicity
* Group B, will receive omeprazole 20 mg, once a day for 12-14 days

Patients will receive treatment for 2~3 weeks during the study, and 2 months of follow up.

Total accrual is anticipated to take 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed exocrine pancreatic cancer with either pathology, histology, or radiology imaging documented as adenocarcinoma
* Patient is a candidate for surgical resection of pancreatic cancer
* ≥ 18 years old at the time of informed consent
* ECOG Performance Status 0-2
* Patients with or without neoadjuvant chemotherapy will be eligible
* Ability to provide written informed consent and HIPAA authorization
* Women of childbearing potential definition must have a negative pregnancy test within 14 days of registration. All women (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) are considered to have childbearing potential unless they meet one of the following criteria:
* Prior hysterectomy or bilateral oophorectomy;
* Has not had menses at any time in the preceding 24 consecutive months
* Candidate for surgery per standard of care of per surgeon's discretion

Exclusion Criteria:

* Patients with pancreatic malignant tumor histologically confirmed as neuroendocrine or any other type of malignancies
* Positive pregnancy test, pregnant, or breastfeeding
* Known hypersensitivity to any component of the formulation or substituted benzimidazoles
* Any other clinically significant laboratory abnormality that would compromise patient safety or the outcome of the study
* Any clinically significant and/or uncontrolled cardiac-related abnormality that would compromise patient safety or the outcome of the study
* Medical condition that might affect the absorption of study medications in the opinion of the investigator.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-07 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Proportion | 2 years
  Proportion of subjects receiving study treatment without adverse events that would significantly delay the surgery
Safety and Tolerability | 2 years
  Frequency and severity of treatment related adverse events per CTCAE v5

SECONDARY OUTCOMES:
v-ATPase LC3-I and LC3-II expression | 2 years
  v-ATPase LC3-I and LC3-II expression on pancreatic tumor
pH | 2 years
  pH of tumor tissue
Correlation | 2 years
  Correlation of biomarker changes with potential cancer cell apoptosis

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Jain, MD, Principal Investigator — University of Oklahoma
Locations (1):
- Stephenson Cancer Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No